CLINICAL TRIAL: NCT05942742
Title: Estimation of Tumor Response With Linac MRI-guided Adaptive Radiotherapy for Locally Advanced Cervical Cancer
Acronym: Gynecolunity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0133
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced Cancer
Keywords: Cervical cancer; Linac MRI; Radiotherapie
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical cancer: Patient treated with Linac MRI for their locally advanced cervical cancer
  Interventions: Device: MRI Linac

INTERVENTIONS:
Device: MRI Linac — External radiotherapy will be performed at Linac MRI, 25 fractions of radiation will be delivered for each patient.The MR-linac offers the ability to individualise and adapt daily treatment plans based on the position or anatomy of the day, following either a simple 'virtual couch shift' adapt-to-position (ATP) approach, or a more complex full reoptimisation adapt-to-shape (ATS) method based on the recontouring of relevant structures. During each radiation therapy, T2-weighted images and diffusion images will be purchased.Treatment plans can be produced and checked by appropriately trained Radiation Oncologists. Each radiation oncologist will decide based on the anatomy of the day the type of workflow to be used (ADP or ATS) for treatment.Patients will undergo accurate image acquisition, registration and interpretation to make sound clinical judgements and proceed to safe and accurate treatment delivery.

SUMMARY:
The management of locally advanced cervical cancer (Figo >IB) is based on radiochemotherapy (RCT) followed by brachytherapy. At present there is no personalized treatment, all patients undergoing radiochemotherapy will follow a conventional treatment by external radiotherapy (46 Gy in 23 sessions associated with cisplatin (CDDP) weekly) and brachytherapy to achieve a total equivalent biological dose around 80-90 Gy).The efficacy of this treatment has been proven for most patients, almost 80% being in complete response after RCT. Nevertheless, on an individual scale, there remains a significant variation in the tumor response, with patients who respond from the first week of treatment, "early responders" or, on the contrary, others who present significant tumor residues after external beam radiotherapy.Various macroscopic tumor volume (GTV) response patterns have been identified based on magnetic resonance imaging (MRI) at diagnosis and MRI before brachytherapy, implying very different clinical target volumes for brachytherapy technique. The difference in tumor volume response has been identified as having a major impact on treatment response.

This is the first study attempting to evaluate tumor response in real time during radiochemotherapy treatment. Knowing the tumor response during treatment will make it possible to modify the management of locally advanced cervical cancer, several therapeutic options might then be discussed depending on the early response to treatment: dose de-escalation for early responders, reduction of time total treatment, personalization of brachytherapy management (technique and dose).

This observational study will allow rapid identification of responder and non-responder patients and might be used as a basis for personalized treatment strategies

ELIGIBILITY:
Inclusion Criteria:

- Women aged ≥ 18 and ≤ 70 years old.

* Histologically confirmed cervical cancer: stage IB2-IVA squamous cell carcinoma or adenocarcinoma (FIGO 2018 criteria), regardless of pelvic lymph node status, no positive lomboaortic lymph nodes. Patients should have no metastatic localization of disease.
* Performance index ≤ 1 (WHO).
* Hematological function: polymorphonuclear neutrophils > 1.5 x 109/L, platelets > 100 x 109/L, hemoglobin > 8,5 g/dL.
* Liver function: total bilirubin < 20 µmol/L or < 12mg/L
* Renal function: creatinine clearance MDRD (Modification of diet in renal disease) >40 ml/min creatinine
* Serum pregnancy test within 7 days before the start of study treatment if risk of pregnancy mentioned by the patient
* Patient able to sign an informed consent form

Exclusion Criteria:

* Previous treatment with radiotherapy, chemotherapy, targeted therapy or immunotherapy treatment for cancer of the cervix or for any other cancer within the previous 5 years.
* Live vaccine, such as yellow fever vaccine.
* History of pelvic irradiation or prior surgical treatment for cancer of the cervix (excluding diagnostic conization).
* Contraindication to MRI imaging (pace maker, metal prosthesis, phobia, etc.)
* Contraindication to the use of cisplatin.
* Inability to perform the follow-up required by the study for geographical, social or psychological reasons.
* History of HIV, HBV or HCV infection with positive serology.
* Pregnant or breastfeeding woman

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible to selection criteria will be included for the next 2 years that is to say 55 patients according to the current active line of patient
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Recist criteria | 8-10 weeks after the end of the treatment
  The local response will be defined by the Recist 1.1 criteria on MRI. The response will be binary, i.e. complete response versus the 3 other categories of the Recist 1.1 classification that is to say partial response, stabilization or progression.
  Nevertheless will identified 3 favorable situation:
  1. complete response on MRI and PET scan
  2. partial response but surgery no performed
  3. partial response, surgery performed and no disease identified on the anatomopathology results

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon-Sud - Radiotherapie/Oncologie, Pierre-Bénite, France